CLINICAL TRIAL: NCT04546139
Title: Feasibility of Smartphone-based Measurement on Badminton Footwork
Status: Completed | Type: Observational
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, YI-JU TSAI, Associate Professor, National Cheng Kung University
Other Study IDs: BadmintonFWApp
Record Dates: First submitted 2020-08-27; First posted 2020-09-11 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fast group
  Interventions: Other: footwork
- slow group
  Interventions: Other: footwork

INTERVENTIONS:
Other: footwork — six-point footwork

SUMMARY:
To evaluate the feasibility of a smartphone-based measurement on badminton footwork. The performance of footwork will be collected utilizing a smartphone app and further investigate the validity, reliability and discrimination of the measurement.

ELIGIBILITY:
Inclusion Criteria:

* adults familiar with badminton six points foot work.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: people who familiar with badminton six points foot work.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
inertial data of footwork performance | a week
  the inertial data collected from both smartphone and IMU sensor during footwork performance. Second assessment was delivered a week after the first assessment

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan